CLINICAL TRIAL: NCT01548508
Title: Evaluation of Functionnal ElectromyoStimulation on Leg In Advanced Chronic Heart Failure After Hospitalisation for Acute Decompensation
Acronym: EMSICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Foundation for the Future, Paris, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0730502; 2008-A00330-55 (Other: Afssaps)
Record Dates: First submitted 2012-02-23; First posted 2012-03-08 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Chronic Heart Failure
Keywords: Advanced Chronic Heart Failure, physical therapy, Exercise
MeSH Terms: conditions — Motor Activity | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functionnal ElectroStimulation (FES) (Experimental)
  Interventions: Other: Functionnal ElectroStimulation (FES)
- SHAM (Sham Comparator)
  Interventions: Other: SHAM

INTERVENTIONS:
Other: Functionnal ElectroStimulation (FES) — Functionnal ElectroStimulation on lower limbs, 1h per day, 5 days per 7, during 6 weeks
  Arms: Functionnal ElectroStimulation (FES)
Other: SHAM — SHAM on lower limbs, 1h per day, 5 days per 7, during 6 weeks
  Arms: SHAM

SUMMARY:
The purpose of the study is to test the efficacy of the Functionnal ElectromyoStimulation (FES) of lower limbs in advanced chronic heart failure. The hypothesis is that FES treatment could improve functional exercise capacity.

DETAILED DESCRIPTION:
Advanced Chronic Heart Failure (ACHF) is a severe and frequent disease inducing a strong limitation of exercise capacity and a poor quality of life. Hospitalisation for cardiac decompensation is frequent and could alter their incapacities because of muscular deconditionning. Tradionnal aerobic rehabilitation exercises fighting against this deconditionning are not relevant in these patients because of dyspnea.

In litterature, Functionnal Electrostimulation (FES) has been tested in stable Chronic Heart Failure (NYHA I to III), far from decompensation. Several authors showed the same improvements than those obtained with conventionnal rehabilitation on aerobic capacities (peak VO2, 6 minutes walking test) and quality of life.

The originality of this study is to test FES soon after acute heart decompensation in ACHF patients. This type of rehabilitation could represent in the future an alternative to conventionnal rehabilitation until the patients could be able to do aerobic exercise.

60 patients will be randomised between two groups, the firsth receiving FES (treatment group), the second receiving skin electrostimulation in the same place without muscular contraction (Sham group). Patient and evaluator do not know what type of stimulation they have. These treatments spread over six weeks, five days per seven. They are began in rehabilitation unit then continued at home.

The principal criteria of judgement of FES efficacy is peak VO2 after the protocol. Secondary criteria are distance to the six minutes walking test, muscular strengh of quadriceps, the muscle mass measured by Dual energy X-ray absorptiometry (DEXA), inflamatory dosage (TNF alpha, IL-1, IL-6, CRP), rest value of Muscle sympathetic nerve activity, score to Minnesota questionnaire and fuctionnal independance.

The attempted results are an significative improvement of aerobic capacity(peak VO2 and six minutes walking test) and the others secondary criteria in FES group compared with Sham group.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Chronic Heart Failure (NYHA III to IV)
* Cardiac Ejection Fraction < 40 %
* peak VO2 < 16 ml/kg/min,
* optimal drug treatment of CHF,
* hospitalised for acute decompensation but not in intensive care

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease with FEV < 50%,
* History of stroke with walking disability, dementia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
VO2 peak | change between baseline and 60 days after the Functional Electromyo Stimulation

SECONDARY OUTCOMES:
Muscle nerve sympathetic activity (MSNA) | change between baseline and 60 days after the Functional Electromyo Stimulation
Six minutes walking test | change between baseline and 60 days after the Functional Electromyo Stimulation
DEXA | change between baseline and 60 days after the Functional Electromyo Stimulation
maximal quadriceps strengh | change between baseline and 60 days after the Functional Electromyo Stimulation
interleukin 1 | change between baseline and 60 days after the Functional Electromyo Stimulation
interleukin 6 | change between baseline and 60 days after the Functional Electromyo Stimulation
TNF alpha | change between baseline and 60 days after the Functional Electromyo Stimulation
CRP | change between baseline and 60 days after the Functional Electromyo Stimulation
BNP | change between baseline and 60 days after the Functional Electromyo Stimulation
score of minessota test | change between baseline and 60 days after the Functional Electromyo Stimulation
score of Functional independency measure | change between baseline and 60 days after the Functional Electromyo Stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Michel GALINIER, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Universty Hospital Toulouse Cardiology, Toulouse, France

REFERENCES:
- [Result] Labrunee M, Despas F, Marque P, Guiraud T, Galinier M, Senard JM, Pathak A. Acute electromyostimulation decreases muscle sympathetic nerve activity in patients with advanced chronic heart failure (EMSICA Study). PLoS One. 2013 Nov 12;8(11):e79438. doi: 10.1371/journal.pone.0079438. eCollection 2013. PMID 24265770